CLINICAL TRIAL: NCT02709551
Title: Comparative Intervention Study of Stress Reduction in Corporate Health Management: Evaluation of the Effects of Heart Rate Variability (HRV) Biofeedback Training, Mindfulness Based Intervention (MBI) and Mindfulness Based HRV-biofeedback
Brief Title: Comparative Intervention Study of Stress Reduction in Corporate Health Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ARCIM Institute Academic Research in Complementary and Integrative Medicine (Other)
Collaborators: Universität Tübingen (Other); Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STM_04
Record Dates: First submitted 2016-02-05; First posted 2016-03-16 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Stress, Psychological
Keywords: corporate health management; hrv; mindfulness
MeSH Terms: conditions — Stress, Psychological

ARMS (3):
- HRV-Bfb (Experimental): HRV biofeedback, training about 30 minutes/day
  Interventions: Behavioral: HRV_Bfb
- MBI (Experimental): Mindfulness based intervention, training about 30 minutes/day
  Interventions: Behavioral: MBI
- MBI_HRV-Bfb (Other): Mindfulness based HRV biofeedback. Wait list control group for the interventions HRV-Bfb and MBI, after the main phase intervention with combined method.
  Interventions: Behavioral: MBI_HRV_Bfb

INTERVENTIONS:
Behavioral: HRV_Bfb
  Arms: HRV-Bfb
Behavioral: MBI
  Arms: MBI
Behavioral: MBI_HRV_Bfb
  Arms: MBI_HRV-Bfb

SUMMARY:
Aim of the study is the evaluation of the effects (psychological and physiological) of an hrv-biofeedback training, a mindfulness training and a combination of both training methods for stress reduction.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* Working in the business in which the study is conducted

Exclusion Criteria:

* Cardiac disease
* Thyroid disease (intake of glucocorticoids)
* Actual psychological illness
* Intake of psychotropic drugs
* Intake of other medication changing HRV

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-02; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Alteration in psychological parameters of stress perception after training | H0: Baseline time point of assessment prior to training H1: Post training time point of assessment (6 weeks after H0) H2: Follow-up (12 weeks after H0) H3: Post training time point of assessment for former wait-list control group (18 weeks after H0)
  We assessed psychological parameters of stress perception with the following questionnaire: TICS ("Trierer Inventar zum chronischen Stress"; Schulz, Schlotz & Becker, 2004). Alteration in data will be statistically compared.
Alteration in psychological parameters of stress coping (behavioral skills) after training | H0: Baseline time point of assessment prior to training H1: Post training time point of assessment (6 weeks after H0) H2: Follow-up (12 weeks after H0) H3: Post training time point of assessment for former wait-list control group (18 weeks after H0)
  We assessed psychological parameters of stress coping with the following questionnaire: SVF 120 ("Stressverarbeitungsfragebogen; Janke & Erdmann, 1997). Alteration in data will be statistically compared.
Alteration in psychological parameters of stress coping (behavior pattern) after training | H0: Baseline time point of assessment prior to training H1: Post training time point of assessment (6 weeks after H0) H2: Follow-up (12 weeks after H0) H3: Post training time point of assessment for former wait-list control group (18 weeks after H0)
  We assessed psychological parameters of stress coping with the following questionnaire: AVEM ("Arbeitsbezogene Verhaltens- und Erlebensmuster"; Schaarschmidt & Fischer, 2008). Alteration in data will be statistically compared.
Alteration in physiological parameters of stress: HRV parameters | H0: Baseline time point of assessment prior to training H1: Post training time point of assessment (6 weeks after H0) H2: Follow-up (12 weeks after H0) H3: Post training time point of assessment for former wait-list control group (18 weeks after H0)
  For the physiological assessment of HRV we used the HRV-Scanner from BioSign GmbH which gathers different HRV parameters like RMSSD and pNN50. HRV was assessed before and after a stressor (Stroop Color-Word Task (based on findings by Stroop, 1935) and D2-R Concentration and Endurance test (Brickenkamp et al., 2010). Alteration in data will be statistically compared.
Alteration in physiological parameters of stress: Salivary cortisol | H0: Baseline time point of assessment prior to training H1: Post training time point of assessment (6 weeks after H0) H2: Follow-up (12 weeks after H0) H3: Post training time point of assessment for former wait-list control group (18 weeks after H0)
  Cortisol was assessed as salivary cortisol (one sample per subject per assessment point). Alteration in data will be statistically compared.

SECONDARY OUTCOMES:
Alteration in psychological parameters of psychological wellbeing after training | H0: Baseline time point of assessment prior to training H1: Post training time point of assessment (6 weeks after H0) H2: Follow-up (12 weeks after H0) H3: Post training time point of assessment for former wait-list control group (18 weeks after H0)
  We assessed psychological wellbeing with the following questionnaire: HEALTH-49 ("Kurzversion der Hamburger Module zur Erfassung allgemeiner Aspekte psychosozialer Gesundheit für die therapeutische Praxis"; Rabung, Harfst, Koch & Schulz, 2007). Alteration in data will be statistically compared.
Alteration in psychological parameters of depression after training | H0: Baseline time point of assessment prior to training H1: Post training time point of assessment (6 weeks after H0) H2: Follow-up (12 weeks after H0) H3: Post training time point of assessment for former wait-list control group (18 weeks after H0)
  We assessed depressive symptoms with the following questionnaire: Beck Depressions-Inventar (BDI-II; Hautzinger, Keller & Kühner; 2006). Alteration in data will be statistically compared.
Alteration in psychological parameters of mindfulness after training | H0: Baseline time point of assessment prior to training H1: Post training time point of assessment (6 weeks after H0) H2: Follow-up (12 weeks after H0) H3: Post training time point of assessment for former wait-list control group (18 weeks after H0)
  We assessed mindfulness with the following questionnaire: FFA 14 ("Kurzversion des Freiburger Fragebogens zur Achtsamkeit"; Walach et al., 2006). Alteration in data will be statistically compared.
Alteration in psychological parameters of self-compassion after training | H0: Baseline time point of assessment prior to training H1: Post training time point of assessment (6 weeks after H0) H2: Follow-up (12 weeks after H0) H3: Post training time point of assessment for former wait-list control group (18 weeks after H0)
  We assessed self-compassion with the following questionnaire: SCS-D-Kurzform ("Self-Compassion Scale"; Hupfeld & Ruffieux, 2011). Alteration in data will be statistically compared.